CLINICAL TRIAL: NCT05224102
Title: A Phase IV, Multicenter, Open-Label, Single-Arm Study to Investigate Faricimab (RO6867461) Treatment Response in Treatment-Naive, Underrepresented Patients With Diabetic Macular Edema
Brief Title: A Study to Investigate Faricimab Treatment Response in Treatment-Naive, Underrepresented Patients With Diabetic Macular Edema
Acronym: ELEVATUM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML43435
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, single-arm study with two phases: the main study phase for all eligible patients (up to 56 weeks), followed by an optional long-term extension phase for eligible patients only in the U.S. (up to 100 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main Phase: Faricimab (Experimental): Participants in the main study phase will receive 6-milligram (mg) faricimab intravitreal (IVT) injections once every 4 weeks (Q4W) up to Week 20, followed by 6-mg IVT faricimab injections once every 8 weeks (Q8W) up to Week 52. Participants will return for the Week 56 safety follow-up visit after ≥28 days following their last study treatment.
  Interventions: Drug: Faricimab
- Long-Term Extension Phase: Faricimab (Experimental): Eligible participants in the U.S. who opt to continue into the long-term extension (LTE) phase of this study will receive 6-mg faricimab IVT injections according to the personalized treatment interval (PTI) dosing algorithm. The minimum and maximum PTIs in the LTE are Q4W and once every 24 weeks (Q24W), respectively.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Participants will receive 6-milligram (mg) faricimab intravitreal (IVT) injections, as described in the study arm descriptions for each study phase.
  Other Names: VABYSMO™; RO6867461; RG7716

SUMMARY:
This study is designed to investigate treatment response in treatment-naïve underrepresented patients with diabetic macular edema (DME) who are treated with faricimab. The study population will consist of participants ≥18 years of age who self-identify as Black/African American, Hispanic/Latino American, or Native American/Alaska Native/Native Hawaiian or other Pacific Islander; in addition, a cohort of Asian Indian participants will be enrolled in India.

ELIGIBILITY:
Inclusion Criteria:

Main Phase General Inclusion Criteria:

* Self-identify as Black/African American, Hispanic/Latino American, or Native American/Alaska Native/Native Hawaiian or other Pacific Islander; or self-identify as Asian Indian residents of the Indian subcontinent
* Diagnosis of diabetes mellitus (type 1 or type 2), as defined by the World Health Organization (WHO) and/or American Diabetes Association, and current regular use of insulin or other injectable drugs (e.g., dulaglutide and liraglutide) and/or oral anti-hyperglycemic agents for the treatment of diabetes
* Hemoglobin A1c (HbA1c) ≤10% (Note: up to 20% of participants enrolled may have HbA1c up to 12%)
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraception methods as defined in the protocol

Main Phase Ocular Inclusion Criteria for Study Eye:

* Intravitreal (IVT) treatment-naïve in the study eye (i.e., have not received previous treatment with any anti-VEGF IVT or any corticosteroids periocular or IVT in the study eye)
* Diabetic macular edema, defined as macular thickening by SD-OCT involving the center of the macula
* BCVA letter score of 73 to 20 letters (both inclusive) using the ETDRS protocol at the initial testing distance of 4 meters at the baseline visit (Day 1)
* Clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images to confirm diagnosis

Long-Term Extension (LTE) Inclusion Criteria:

* Enrollment in and completion of the main study, without discontinuation from study or study drug treatment
* Signed LTE-phase Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraception methods as defined in the protocol

Exclusion Criteria:

Main Phase General Exclusion Criteria:

* Diabetes mellitus (type 1 or type 2) that is currently medically untreated
* Previously untreated diabetes mellitus (type 1 or type 2) who started on oral or injectable anti-diabetic medication within 3 months prior to Day 1
* Any known hypersensitivity to any of the components in the faricimab injection
* Any known hypersensitivity to any contrast media (e.g., fluorescein), dilating eye drops, disinfectants (e.g., iodine), or any of the anesthetics and antimicrobial preparations used by the patient during the study
* History of other diseases, other non-diabetic metabolic dysfunction, physical examination finding, or historical or current clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of the faricimab or that might affect interpretation of the results of the study or renders the patient at high-risk for treatment complications, in the opinion of the investigator
* Active cancer within the past 12 months prior to Day 1 except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤6 and a stable prostate-specific antigen for >12 months
* Stroke (cerebral vascular accident) or myocardial infarction within 12 months prior to Day 1
* Any febrile illness within 1 week prior to Day 1
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of faricimab
* Uncontrolled blood pressure, defined as systolic >180 mmHg and/or diastolic >100 mmHg (while patient is at rest in a sitting position); if a patient's initial reading exceeds these values, a second reading may be taken ≥30 minutes later on the same day
* Renal failure requiring renal transplant, hemodialysis, or peritoneal dialysis within 6 months prior to Day 1 or anticipated to require hemodialysis or peritoneal dialysis at any time during the study
* Any condition resulting in a compromised immune system that is likely to impact the aqueous humor inflammatory biomarkers
* Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins or minerals) within 3 months (or 5 half-lives, whichever is longer) prior to Day 1, or during the course of this study
* Substance abuse occurring within 12 months prior to screening, in the investigator's judgment
* Use of systemic immunomodulatory treatments (e.g., IL-6 inhibitors) within 6 months or 5 half-lives (whichever is longer) prior to Day 1
* Use of any systemic corticosteroids within 1 month prior to Day 1
* Systemic treatment for suspected or active systemic infection
* Any prior or concomitant systemic anti-VEGF treatment within 6 months or 5 half-lives (whichever is longer) prior to Day 1
* Use of systemic medications known to be toxic to the lens, retina, or optic nerve (e.g., deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines, or ethambutol) during the 6-months (or 5 half-lives, whichever is longer) prior to Day 1
* Receiving any treatment that leads to immunosuppression within 6 months (or 5 half-lives, whichever is longer) prior to Day 1
* Requiring continuous use of any medications or treatments listed as prohibited therapy

Main Phase Ocular Exclusion Criteria for Study Eye:

* High-risk proliferative diabetic retinopathy (PDR) in the study eye, using any of the following established criteria for high-risk PDR: Any vitreous or pre-retinal hemorrhage; Neovascularization elsewhere ≥1/2 disc area within an area equivalent to the mydriatic ETDRS 7 or 4 fields on clinical examination or on CFPs; Neovascularization at disc ≥1/3 disc area on clinical examination
* Tractional retinal detachment, pre-retinal fibrosis, vitreomacular traction, or epiretinal membrane involving the fovea or disrupting the macular architecture in the study eye, as evaluated by the central reading center
* Any history of or ongoing rubeosis iridis
* Any panretinal photocoagulation or macular laser (focal, grid or micropulse) photocoagulation treatment received in the study eye prior Day 1
* Any history of treatment with anti-VEGF or any periocular or IVT corticosteroids in the study eye prior to Day 1
* Any treatment for dry eye disease in the last month prior to Day 1 (e.g., cyclosporine eye drops, lifitegrast eye drops). Lubricating eye drops and ointments are permitted.
* Any treatment with anti-inflammatory eye drops (e.g., doxycycline) within 1 month prior to Day 1
* Any intraocular surgery (e.g., cataract surgery) within 3 months prior to Day 1 or any planned surgery during the study
* Any glaucoma surgery prior to the screening visit
* History of vitreoretinal surgery/pars plana vitrectomy, corneal transplant, or radiotherapy
* Uncontrolled glaucoma
* Any active or suspected ocular or periocular infections on Day 1
* Any presence of active intraocular inflammation on Day 1 (i.e., Standardization of Uveitis Nomenclature [SUN] criteria >0 or National Eye Institute [NEI] vitreous haze grading >0) or any history of intraocular inflammation
* Any history of idiopathic, infectious, or noninfectious uveitis
* Any current ocular condition or other causes of visual impairment for which, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema

Main Phase Ocular Exclusion Criteria for Non-Study Eye:

* Any history of idiopathic or immune-mediated uveitis
* Active ocular inflammation or suspected or active ocular or periocular infection on Day 1
* Currently receiving treatment with brolucizumab or bevacizumab in the non-study eye and is unwilling to switch to a protocol-allowed, non-study eye anti-VEGF treatment during the study
* Any previous treatment with Iluvien® or Retisert® (fluocinolone acetonide IVT implant) in the non-study eye
* Non-functioning non-study eye, defined as either: BCVA of hand motion or worse; No physical presence of non-study eye (i.e., monocular); or, Legally blind in the patient's relevant jurisdiction

Long-Term Extension (LTE) Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final IVT injection of faricimab
* Presence of other ocular diseases that give reasonable suspicion of a disease or condition that contraindicates the use of faricimab, that might affect interpretation of the results of the LTE, or that renders the patient at high risk for treatment complications
* Presence of other diseases, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of faricimab and that might affect interpretation of the results of the LTE, or that renders the patient at high risk of treatment complications
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab injections, study treatment procedure, dilating drops, or any of the anesthetic and antimicrobial preparations used by a patient during the LTE phase
* Requirement for continuous use of any medications or treatments indicated as prohibited therapy (as defined in the protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Main Phase: Change in Best Corrected Visual Acuity (BCVA) from Baseline at Week 56, as Measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart at a Starting Distance of 4 Meters | From Baseline to Week 56
Long-Term Extension Phase: Incidence and Severity of Ocular Adverse Events | From Day 1 until end of long-term extension (up to 100 weeks)
Long-Term Extension Phase: Incidence and Severity of Non-Ocular Adverse Events | From Day 1 until end of long-term extension (up to 100 weeks)

SECONDARY OUTCOMES:
Main Phase: Percentage of Participants with a Greater Than or Equal to (≥)2-Step ETDRS Diabetic Retinopathy Severity Scale (DRSS) Improvement from Baseline Over Time | Baseline and Weeks 20 and 56
Main Phase: Percentage of Participants with a ≥3-Step ETDRS Diabetic Retinopathy Severity Scale (DRSS) Improvement from Baseline Over Time | Baseline and Weeks 20 and 56
Main Phase: Percentage of Participants with Absence of Intraretinal Fluid Over Time | Baseline and Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, 52, and 56
Main Phase: Percentage of Participants with Absence of Subretinal Fluid Over Time | Baseline and Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, 52, and 56
Main Phase: Change from Baseline in Central Subfield Thickness Over Time | Baseline and Weeks 4, 8, 12, 16, 20, 28, 36, 44, 48, 52, and 56
Main Phase: Percentage of Participants Gaining ≥15 or ≥10 Letters in BCVA from Baseline at Week 56 | Baseline and Week 56
Main Phase: Percentage of Participants Avoiding a Loss of ≥15 or ≥10 Letters in BCVA from Baseline at Week 56 | Baseline and Week 56
Main Phase: Incidence and Severity of Ocular Adverse Events | From Baseline up to Week 56
Main Phase: Incidence and Severity of Non-Ocular Adverse Events | From Baseline up to Week 56
Main Phase: Number of Participants Testing Positive for Anti-Drug Antibodies (ADAs) Against Faricimab at Baseline and Anytime During the Study | From Baseline up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (43):
- United States (33):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Win Retina, Arcadia, California
  - Retinal Diagnostic Center, Campbell, California
  - Retina Consultants of Orange County, Fullerton, California
  - Kaiser Permanente Southern California, Los Angeles, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Southwest Retina Consultants, Durango, Colorado
  - Emerson Clinical Research Institute LLC, Washington D.C., District of Columbia
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Retina Macula Specialists of Miami - LeJeune Road Office, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Wilmer Eye Institute Johns Hopkins University, Baltimore, Maryland
  - Md Medical Research, Oxon Hill, Maryland
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Retina Consultants of Nevada, Henderson, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - The Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina - Teaneck, Teaneck, New Jersey
  - Piedmont Retina Specialists, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, INC, Beachwood, Ohio
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Memphis, Tennessee
  - Austin Clinical Research LLC, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Brown Retina Institute, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
- India (7):
  - MM Joshi Eye Institute, Hubli, Karnataka
  - PBMA'S H. V. Desai Eye Hospital, Pune, Maharashtra
  - M & J Western Regional Institute of Ophthalmology, Ahmedabad, Rajasthan
  - Sankara Nethralaya, Chennai, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Regional Institute of Ophthalmology, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
- Kenya (2):
  - Nairobi Hospital, Nairobi
  - City Eye Hospital, Nairobi
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No